CLINICAL TRIAL: NCT02646046
Title: A Study of Evaluation of Effectiveness on the Combining Performance of Call Emergency Medical System (EMS) and Simultaneous Chest Compressions With One Hand in a Lone Rescuer CPR: a Simulation Study Using the Manikin
Brief Title: Combining Performance of Call EMS and Simultaneous Chest Compressions in a Lone Rescuer CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Assistant Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CallplusCPR
Record Dates: First submitted 2015-12-23; First posted 2016-01-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Cardiopulmonary Resuscitation; Emergency Medical Services; Cell phones; Simulation Training
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combi lone-CPR (Experimental): Intervention group
  : Newly developed method
  Interventions: Behavioral: Combi lone-CPR
- Conventional lone-CPR (Active Comparator): Conventional CPR group
  Interventions: Behavioral: Conventional lone-CPR

INTERVENTIONS:
Behavioral: Combi lone-CPR — When study participants meet the arrest victim (simulated), they start chest compression and call for help to EMS at the same time, then continue the chest compression and 2 breath alternatively until the EMS arrival
  Arms: Combi lone-CPR
Behavioral: Conventional lone-CPR — When study participants meet the arrest victim (simulated), they first call for help to EMS and then start chest compression and 2 breath alternatively until the EMS arrival
  Arms: Conventional lone-CPR

SUMMARY:
Investigators designed the novel combining technique that rescuer start the chest compression with one hand during calling for help to the Emergency Medical System (EMS) via a cell phone with another hand when he witnessed the arrest victim. This method may be helpful to reduce the hand-off time and increase the faction time of chest compression until the arrival of EMS members.

To verify this hypothesis, we conducted a random, controlled simulation study.

DETAILED DESCRIPTION:
This study used a random, controlled design in the simulation setting using a manikin. Study participants were recruited from healthy adult (age > 18 years) laypersons who attended the BLS training courses provided by the BLS training class.

The simulation scenario consists of witness of an out of hospital cardiac arrest and activation of the EMS system with the prepared cellular phone. Interventional method contained the immediate starting of the chest compression with one hand during the calling for help to the EMS via a cell phone with another hand.

We compare the quality of CPR between the novel interventional method (start CPR during Call to EMS) and conventional method (First Call to EMS and then start CPR).

ELIGIBILITY:
Inclusion Criteria:

* All healthy volunteers who attended the basic CPR training class
* Agreement with the simulation trial

Exclusion Criteria:

* volunteers who had some healthy problem which may affect the study results
* Not agreement with the simulation trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Total numbers of chest compression with correct depth | 3 minutes
  correct depth is defined as depth > 50 mm

SECONDARY OUTCOMES:
Incomplete release of chest compression | 3 minutes
Incorrect position of chest compression | 3 minutes
Correct Tidal volume | 3 minute
  defined as 500-800 ml in manikin setting
Interruption time of chest compression | 3 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koster RW, Baubin MA, Bossaert LL, Caballero A, Cassan P, Castren M, Granja C, Handley AJ, Monsieurs KG, Perkins GD, Raffay V, Sandroni C. European Resuscitation Council Guidelines for Resuscitation 2010 Section 2. Adult basic life support and use of automated external defibrillators. Resuscitation. 2010 Oct;81(10):1277-92. doi: 10.1016/j.resuscitation.2010.08.009. No abstract available. PMID 20956051
- [Background] Berg RA, Hemphill R, Abella BS, Aufderheide TP, Cave DM, Hazinski MF, Lerner EB, Rea TD, Sayre MR, Swor RA. Part 5: adult basic life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S685-705. doi: 10.1161/CIRCULATIONAHA.110.970939. PMID 20956221
- [Background] Riera SQ, Gonzalez BS, Alvarez JT, Fernandez Mdel M, Saura JM. The physiological effect on rescuers of doing 2min of uninterrupted chest compressions. Resuscitation. 2007 Jul;74(1):108-12. doi: 10.1016/j.resuscitation.2006.10.031. Epub 2007 Feb 14. PMID 17303308